CLINICAL TRIAL: NCT06678061
Title: Efficacy of Radiofrequency Splanchnic Denervation Compared to Neurolytic Retrocrural Celiac Plexus Block for Patients with Chronic Upper Abdominal Cancer Pain
Brief Title: Radiofrequency Splanchnic Denervation ,neurolytic Retrocrural Celiac Plexus Block Chronic Upper Abdominal Cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, NourhanMohammedAlaaElgalaly, PRINCIPLE INVESTIGATOR, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERSDCNRCPBPCUACP
Record Dates: First submitted 2024-11-04; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- radiofrequency splanchnic denervation (Active Comparator): Radiofrequency ablation of splenic nerve. The nerves were then anesthetized with 2 mL of 2% lidocaine before RF performed. In RFA group, lesion will be performed at 80 degrees celsius for 3 lesions 2 minutes each on both sides.
  Interventions: Device: radiofrequency
- Celiac plexuc block (Active Comparator): Neurolytic ablation of the celiac plexus.Two milliliter of contrast material will be injected in each side for confirmation a test injection with 5 mL of 2% lidocaine to both sides, and wait for 5 minutes then inject 5 ml of 100% alcohol will in each side after 5 minutes to allow the local anesthetic to take action. 1 ml of 2%
  Interventions: Device: radiofrequency

INTERVENTIONS:
Device: radiofrequency — block of neurolytic retrocrural celiac plexus block
  Other Names: plexus block

SUMMARY:
To compare between the efficacy of radiofrequency splanchnic denervation and neurolytic retrocrural celiac plexus block in chronic upper abdominal cancer pain

DETAILED DESCRIPTION:
Abdominal cancers are not uncommon, according to WHO latest updates in cancer epidemiology published in 2020, the percentage of new cases incidence is rapidly increasing as follow: Colon (6.0%), Stomach (5.6%), Liver (4.7%), Esophagus (3.1%), Pancreas (2.6%), and Gall bladder (0.6%).

Pain is one of the chief complains in cancer patients and the leading cause for seeking medical advice. In abdominal malignancies, visceral pain is poorly localized due to both fewer receptors participating in the process of visceral pain and the scarce representation within the primary somatosensory cortex. The challenge in identifying the pain generators and effectively treat this condition explains the tendency for abdominal pain to become chronic and frustration associated with its management for both the patient and the health care provider. Effective analgesia has become sometimes difficult to institute in abdominal cancer patients because the dose-response is unpredictable and the analgesic doses may be poorly tolerated in patients who are debilitated and using several other drugs as they are usually old age, complaining of nausea, repeated vomiting, and dehydration, elevated liver enzymes especially in liver affection by primary or secondary lesions.

Many patients may have residual symptoms that impact their quality of life despite thoughtful pharmacologic and surgical treatment. So, Non pharmacologic strategies, including physical therapy, integrated and complementary medicine, lifestyle modifications, and interventional procedures may also be useful adjuncts to surgical and pharmacologic therapy.

Thus, the neurolytic sympathetic block has been proposed as an efficient, relatively simple, and repeatable method of management, bringing both relief of pain and allowing the discontinuation of drugs or at least a decrease in their dosage.

Frequently used nerve ablation and modulation methods include conventional radiofrequency ablation (RFA) using heat and chemical ablation using alcohol.

The celiac plexus lies anterior to aorta at the level of the first lumber vertebra. A block of the celiac plexus is applied most commonly to patients with pancreatic, gastric, or biliary cancer, as such patients typically have severe intractable upper abdominal pain . Splanchnic nerves are paired nerves arising from the thoracic sympathetic trunk (ganglia 5 to 12) which pierce the crura of the diaphragm at the T11 and T12 levels to join the celiac ganglion. Interruption of these nerve fibers can provide relief from pain associated with intra-abdominal malignancies .Neurolysis reduces pain by disrupting pain signals along the neural pathway The celiac plexus and splanchnic nerves are targets for neurolytic blocks for pain relief from pain caused by upper gastrointestinal tumors. And in this trial we are aiming to compare between the efficacies of both techniques in the management of chronic upper abdominal cancer pain.

:

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged from 20-70 years old, with upper GIT tumors, including cancer of the lower third of the esophagus, stomach cancer, pancreatic cancer, cancer liver, and cancer of the biliary tract,
2. Abdominal cancer pain: includes patients with NRS pain score ≥ 5. [16]
3. Included participants should show adequate response to diagnostic block for the splanchnic nerves, i.e. reduction of NRS pain score > 50% at least for 2 hours

Exclusion Criteria:

- a- Patient's refusal. b- Patients medical condition as: coagulopathies, moderate or major cardiac/respiratory incapacitating diseases, liver or renal failure, infection either systemic or localized and anatomical anomalies or lesions at the spine.

c- Any psychiatric illness that would interfere with the perception and the assessment of pain, and any reason that would result in the protocol violation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
the Numeric Pain Rating Scale (NRS) pain scale | 6 months
  Change in the Numeric Pain Rating Scale (NRS) pain scale at the first 2 weeks compared to the pre-procedural pain

SECONDARY OUTCOMES:
1- Total opioid consumption | 6 months
  daily consumption of opioid
Functional Assessment of Chronic Illness Therapy or Cancer Therapy (FACT) | 6 months
  measure patient quality of life
Patient Health Questionnaire (PHQ-9) | 6 months
  measure depression and anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Samy Erfan, MD, Study Director — AssiutUniversity; Nourhan Elgallay, Msc, Principal Investigator — Assiut University
Locations (2):
- Egypt (2):
  - Assiut University, Asyut, Asyut Governorate
  - South Egypt Cancer Institute, Asyut, Asyut Governorate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilbody S, Richards D, Brealey S, Hewitt C. Screening for depression in medical settings with the Patient Health Questionnaire (PHQ): a diagnostic meta-analysis. J Gen Intern Med. 2007 Nov;22(11):1596-602. doi: 10.1007/s11606-007-0333-y. Epub 2007 Sep 14. PMID 17874169
- [Background] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841
- [Background] Cherny N, Ripamonti C, Pereira J, Davis C, Fallon M, McQuay H, Mercadante S, Pasternak G, Ventafridda V; Expert Working Group of the European Association of Palliative Care Network. Strategies to manage the adverse effects of oral morphine: an evidence-based report. J Clin Oncol. 2001 May 1;19(9):2542-54. doi: 10.1200/JCO.2001.19.9.2542. PMID 11331334
- [Background] Miguel R. Interventional treatment of cancer pain: the fourth step in the World Health Organization analgesic ladder? Cancer Control. 2000 Mar-Apr;7(2):149-56. doi: 10.1177/107327480000700205. PMID 10783819
- [Background] Peipert JD, Cella D. Bifactor analysis confirmation of the factorial structure of the Functional Assessment of Cancer Therapy-General (FACT-G). Psychooncology. 2019 May;28(5):1149-1152. doi: 10.1002/pon.5062. Epub 2019 Apr 17. No abstract available. PMID 30883962
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359